CLINICAL TRIAL: NCT02835404
Title: A Randomized, Open Label, Single Centre Clinical Trial of Pelvic External Radiotherapy Combined With 252-Cf Neutron Intracavitary Brachytherapy With or Without Platinum in Treatment of Local Advanced Cervical Cancer
Brief Title: Pelvic External Combined With 252-Cf Neutron Intracavitary Radiotherapy With or Without Platinum in Treating Advanced Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Xin Lei, M.D.Prof, M.D, Prof., Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012012
Record Dates: First submitted 2016-07-06; First posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-06

CONDITIONS: Cervical Cancer; Complications
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — nedaplatin

ARMS (2):
- Concurrent radiochemotherapy Group (Experimental): Concurrent radiochemotherapy with Nedaplatin Pelvic External Radiotherapy: patients received 20 Gy2.0/f, for 25-27f with 8mv-X rays (SSD) 252-Cf Neutron Intracavitary Brachytherapy: total dose of reference point A was 4400cGy, in four times Transvaginal implant sessions during Pelvic External Radiations; Chemotherapy: Nedaplatin(NDP) 30-40mg/m2 iv., on day1, 4weeks as one cycle
  Interventions: Drug: Nedaplatin; Radiation: Pelvic External Radiotherapy; Radiation: 252-Cf Neutron Intracavitary Brachytherapy
- Radiotherapy Group (Active Comparator): patients received Radiotherapy only Pelvic External Radiotherapy: patients received 20 Gy2.0/f, for 25-27f (SSD)with 8mv-X Linear Accelerator SSD 252-Cf Neutron Intracavitary Brachytherapy: total dose of reference point A was 4400cGy, in four times Transvaginal implant sessions during Pelvic External Radiations.
  Interventions: Radiation: Pelvic External Radiotherapy; Radiation: 252-Cf Neutron Intracavitary Brachytherapy

INTERVENTIONS:
Drug: Nedaplatin — Chemotherapy: Nedaplatin(NDP) 30-40mg/m2 iv., on day1, 4weeks as one cycle
  Other Names: NDP
  Arms: Concurrent radiochemotherapy Group
Radiation: Pelvic External Radiotherapy — patients received 20 Gy2.0/f, for 25-27f (SSD)with 8mv-X rays (SSD)
Radiation: 252-Cf Neutron Intracavitary Brachytherapy — total dose of reference point A was 4400cGy, in four times Transvaginal implant sessions during Pelvic External Radiations

SUMMARY:
The objective of this study was to evaluate the efficacy and complication of the treatment of pelvic external combined with 252-Cf neutron intracavitary radiotherapy with or without platinum in local advanced cervical cancer patients in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* 1. To be aged from 18 (including 18) to 65 (including 65), female patient;
* 2. Expected survival ≥6 months
* 3. Pathologically proven diagnosis of squamous carcinoma or adenocarcinoma of the cervix, according to FIGO(International Federation of Gynecology and Obstetrics) staging, appropriate stage for protocol entry, including IIA2, IIB,IIIA,IIIB;
* 4. No patients with distant metastases;
* 5. Measurable target lesions (satisfying the criteria in RECIST 1.1);
* 6. ECOG PS status of 0-2;
* 7. No prior treatment;
* 8. No
* 9. No surgery
* 10. Major organ function has to meet the following criteria:

  1. Bilirubin <1.5 times the upper limit of normal (ULN)
  2. ALT , AST and APL≤2.5 × ULN
  3. NEUT≥2.0 × 10^9 / L
  4. PLT ≥ 100 × 10^9 / L
  5. HB≥60g/L
  6. Serum Cr and urea nitrogen ≤ 1.5 × ULN
* 11. Favorable cardiac functions, no patients with myocardial infarction within half a year, hypertension and coronary disease are well-controlled.

Exclusion Criteria:

* 1. Serious heart disease, pulmonary disease, hepatic disease, , renal disease and metabolic disease, or with electrolyte disturbance;
* 2. Allergic to platinum;
* 3. Rejecte to join the study in other conditions.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-06 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity events | Week 5 of Radiation Therapy (RT)
  chemo-related toxicity as measured by CTCAE v. 4.0, radiation-related toxicity as measured by RTOG/EORTC criteria
Long-trem toxicity events | through study completion, an average of 5 year
  chemo-related toxicity as measured by CTCAE v. 4.0, radiation-related toxicity as measured by RTOG/EORTC criteria

SECONDARY OUTCOMES:
2 Years Overall survial Rate | 2 years
  chemo-related toxicity as measured by CTCAE v. 4.0, radiation-related toxicity
3 Years Overall survial Rate | 3 years
5 Years Overall survial Rate | 5 years
Disease-free survival (DFS) | through study completion, an average of 3 year
Overall survial (OS) | through study completion, an average of 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lei, M.D, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, China